CLINICAL TRIAL: NCT04248764
Title: Investigating the Effects of Different Soft Tissue Mobilizations on Delayed Onset Muscle Soreness and Performance in Recreational Athletes: A Single Blinded, Randomized Controlled Study
Brief Title: Investigating the Effects of Different Soft Tissue Mobilizations on Delayed Onset Muscle Soreness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Katip Celebi University (Other)
Responsible Party: Principal Investigator, Umut Ziya Kocak, Research Assisstant, Izmir Katip Celebi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2019-KAE-0372
Record Dates: First submitted 2020-01-27; First posted 2020-01-30 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: Muscle Soreness
Keywords: Recreational athlete; Soft Tissue Mobilization; Delayed Onset Muscle Soreness
MeSH Terms: conditions — Myalgia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Foam roller group (Experimental): Participants will perform a 100 fall-bounces (5 sets x 20 reps, with two minutes of rest) from a 50 cm high box as the fatigue protocol. All participants will use a five-minute bicycle ergometer to warm up prior to the. Following the fatigue protocol, foam roler will be applied to the participants' quadriceps femoris muscles in a prone position for five minutes.
  Interventions: Other: Foam roller application
- Massage group (Experimental): Participants will perform a 100 fall-bounces (5 sets x 20 reps, with two minutes of rest) from a 50 cm high box as the fatigue protocol. All participants will use a five-minute bicycle ergometer to warm up prior to the. Following the fatigue protocol, sports massage will be applied on the quadriceps femoris muscles for five minutes.
  Interventions: Other: Massage application
- Control group (No Intervention): Participants will perform a 100 fall-bounces (5 sets x 20 reps, with two minutes of rest) from a 50 cm high box as the fatigue protocol. All participants will use a five-minute bicycle ergometer to warm up prior to the. Following the fatigue protocol, the participants will rest in the long sitting position for 5 minutes.

INTERVENTIONS:
Other: Foam roller application — Following the fatigue protocol, foam roller application will be applied to the quadriceps femoris muscle for five minutes in the prone position.
  Arms: Foam roller group
Other: Massage application — Following the fatigue protocol, sports massage will be applied to the quadriceps femoris muscle for five minutes.
  Arms: Massage group

SUMMARY:
Delayed onset muscle soreness (DOMS) is associated with the initiation of a new physical activity or a sudden increase in exercise volume and intensity. DOMS also occurs following eccentric exercises such as ballistic stretching, downhill running, weight training and plyometrics. DOMS might prevent performing sports and decreases the performance of professional or recreational athletes. Recently, different soft tissue mobilization applications (massage, foam roller) have been preferred by many athletes to prevent DOMS. However, there is no study comparing the effects of these techniques on DOMS. Therefore, the aim of the present study is to investigate the effects of different soft tissue mobilization practices on DOMS and sportive performance in recreational athletes. In order to achieve this goal, a total of 36 recreational athletes will be included and will be allocated to three groups as foam roller group (n=12), massage group (n=12) and control group (n=12). Demographic data, thermal camera measurements, fatigue level assessments, and performance measurements will be performed. All measurements will be carried out four times as before the application, immediately after the application, after 24 hours and after 48 hours.

DETAILED DESCRIPTION:
After being invited to the study, the demographic data of all participants who agreed to participate in the study will be recorded on a structured form. Participants will be randomly divided into three groups: Massage application group, Foam Roller application group and Control group. Afterwards, thermal imaging, perceived fatigue and pain level, blood lactate level measurements, and vertical jump assessments will be done for the quadriceps femoris muscle. Then, the fatigue protocol will be applied for the quadriceps femoris muscle and five-minute applications will be made according to the groups in which they are randomly separated. Evaluations made in the first applications will be made immediately after the applications, 24 hours and 48 hours later, as the 2nd, 3rd and 4th measurements. The assessor will not know which group the participants are from.

ELIGIBILITY:
Inclusion Criteria:

* Performing recreational sports at least 1 and at most 3 times a week.

Exclusion Criteria:

* Any musculoskeletal, neurological or other serious health problems experienced in the past six months
* Not willing to participate in the study

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2021-02-10 (Actual); Primary Completion 2023-01-30 (Actual); Study Completion 2023-03-14 (Actual)

PRIMARY OUTCOMES:
Tissue Temperature Change | Four measurements will be performed as immediately before, immediately after, 24 hours and 48 hours later from fatigue protocol.
  Tissue temperature change will be assessed by using thermal camera imaging which is a non-invasive method. By determining the temperature differences in the tissues with the thermal camera, it will be determined in which regions the circulation increases or decreases.
Blood Lactate Level Change | Four measurements will be performed as immediately before, immediately after, 24 hours and 48 hours later from fatigue protocol.
  Lactate Edge will be used and the lactate levels will be measured from a drop of blood.

SECONDARY OUTCOMES:
Perceived Fatigue and Pain Level Changes | Four measurements will be performed as immediately before, immediately after, 24 hours and 48 hours later from fatigue protocol.
  By using a 0-100 millimeter visual analog scale (0: none, 100: maximum), the participants will determine the fatigue and pain levels. Higher scores indicate worse fatigue and pain.
Change in Lower Extremity Anaerobic Performance | Four measurements will be performed as immediately before, immediately after, 24 hours and 48 hours later from fatigue protocol.
  Vertical jump test will be used to evaluate the lower extremity anaerobic performance.

CONTACTS AND LOCATIONS:
Overall Officials: Umut Ziya Kocak, Study Director — Izmir Katip Celebi University
Locations (1):
- Izmir Katip Celebi University, Izmir, Turkey (Türkiye)